CLINICAL TRIAL: NCT00832676
Title: Exploring the Learning Needs of Individuals With Inflammatory Arthritis From the Perspectives of Patients, Family Members and Friends, and Health Care Providers: Patient Perspectives (Focus Groups)
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Dr. Mary J. Bell, Sunnybrook Health Sciences Centre
Other Study IDs: DOCH2 447-2008
Record Dates: First submitted 2009-01-26; First posted 2009-01-30 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Arthritis
Keywords: Mixed methods research (qualitative and quantitative); Peer support; Early inflammatory arthritis; Self-management; Patient education
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Inflammatory arthritis (IA) is a major cause of long-term disability. Due to specialist shortages, failure of primary care providers and individuals to recognize the disease, and lack of awareness of the importance of early intervention, delays to rheumatologic care are common. Peer support models have been used for various health issues and may be one method to assist individuals with early IA to manage their disease and cope with stress. Qualitative research methods (focus groups) will seek out feedback on a peer support approach and explore the learning needs (informational needs, educational preferences) and opinions about emotional and appraisal support of individuals living with IA, from the perspectives of patients. The data will be analyzed and expressed themes (articulated needs and understandings of interviewee context) will guide the future development of a peer support intervention.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL

____________________________________________________________________

Exploring the Learning Needs of Individuals with Inflammatory Arthritis from the Perspectives of Patients, Family Members and Friends, and Health Care Providers: Patient Perspectives

_____________________________________________________________________

RATIONALE

Rheumatic diseases are a chronic, lifelong illness that results in significant pain, disability, and morbidity in the Canadian population (Perruccio, Power & Badley, 2006). Focusing on one aspect of rheumatic diseases, inflammatory arthritis has been associated not only with the aforementioned concerns, but also with an increased burden of care that affects not only patients, but extends its impact to include their family members, friends, and caregivers. Inflammatory arthritis is also associated with significant increases to healthcare budgets (Hunsche, Chancellor & Bruce, 2001). Care and management of these diseases are expected to be in high demand as the burden of illness is estimated to be on the rise (Perruccio, Power & Badley, 2006). The number of primary care providers and specialists is not sufficient to meet this anticipated increase, (Beaulieu et al., 2004; Glazier et al., 2003) and patients dealing with chronic diseases are increasingly required to self-manage their disease. This can be a stressful and daunting process for a newly diagnosed patient and may result in delayed decision-making and ultimately, delays in their disease treatment.

While physician care is undeniably important in the management of inflammatory arthritis, educating patients with the knowledge and skills to self-manage their disease can be helpful with decision-making processes and reducing healthcare burden. For example, Lorig et al (2001) demonstrated that individuals who were better able to self-manage their illness experienced a significant improvement in health behaviours, self-efficacy, and health status, and had fewer visits to emergency departments. By equipping patients with strategies to cope and enhance personal health, they take on a more active role in the management of their disease and are able to take on health promoting activities with little supervision from healthcare professionals (Keysor et al., 2003). In fact, patient education in self-management has been identified as an arthritis best-practice and a key clinical practice guideline and (Combe et al., 2007; Holbrook, 2000; Jordan et al., 2003).

Patient education can take many forms, but peer support interventions have been particularly effective in helping patients manage chronic diseases, including HIV, alcoholism and diabetes. Likewise, we hope to examine the benefits, challenges, and impact peer support can have on individuals living with inflammatory arthritis. A peer is someone who shares a common characteristic, such as age, gender, social economic status, education, religion, or in this case, status of disease (Doull et al., 2005). Peers have experiential knowledge of rheumatic disease, its management and care, and the social implications it has had in their lives. Within a healthcare context, they can provide assistance to individuals living with arthritis by providing support to their emotional, appraisal, and informational needs. Peers have the potential to influence health outcomes of other patients by addressing feelings of isolation and loneliness, promoting positive outlook and motivation, and providing information about behaviors that encourage health and well-being (Dennis, 2003). They can augment the services provided by healthcare professionals and can help individuals with inflammatory arthritis better cope and manage their illness. While peer support groups have been used to address many chronic diseases, their implementation amongst individuals with inflammatory arthritis has been limited. The effectiveness of such a program is dependent on the educational preferences and learning needs of its participants and this is a topic that requires examination and further assessment.

PURPOSE AND OBJECTIVE

This project addresses one subcomponent of a larger study in which the overall purpose is to explore the learning needs (informational needs, emotional needs, and appraisal needs) and the educational preferences of individuals with inflammatory arthritis. The impact of formal or informal peer support on individuals with rheumatic disease and the improvement of their health and well-being will also be examined with an emphasis on peer support from the perspective of patients living with the disease.

This project will focus on soliciting perspectives of patients with inflammatory arthritis. To better understand the learning needs and potential impact of peer support strategies, including the context, circumstances, and processes involved in making peer support an effective intervention. This project, in particular, will examine:

* the perspective of individuals with inflammatory arthritis regarding disease management and educational needs
* what they feel are their emotional, informational, appraisal needs
* what specific feedback they are seeking related to peer support
* whether and how these needs change over the progression and duration of the disease course

METHODOLOGY

Qualitative examination of the aforementioned objectives will be carried out using focus groups.

Study Design

Eligible study participants will be divided into three focus groups of 6-8 participants each based on their disease duration:

* 0-6 months
* Over 6 months - 2 years
* 2 - 5 years

Each focus group will be comprised of individuals with inflammatory disease of mixed age and gender. Focus group sessions will be held over several weeks and at a time convenient to the participants. This will be done in order to avoid conflicts with work and shift schedules. Informed, written consent will also be obtained from potential participants (Appendix 1 - Information Sheet and Appendix 2 - Consent Form).

Two second-year medical student co-investigators and/or the study coordinator from the University of Toronto will be present at each focus group session. A semi-structured interview guide will be used (Appendix 3 - Interview Guide) with probes to prompt further discussion when appropriate. One medical student will conduct the focus group while the second student or study coordinator will keep a speaker log and take notes throughout the session. Each participant will be assigned a number and a record will be kept of the first phrase of each speaker. The speaker log will be used to aid in the analysis (i.e. to clarify if the view was expressed by a number of people or one person many times). During focus group discussions, only the first name of each participant will be used.

Focus group sessions will run approximately 1 ½ - 2 hours in duration. After every session, each medical student/study coordinator will create field notes in which they will independently record their thoughts and impressions of the interview, non-verbal communication, and other conversations not recorded before or after the meeting. Each focus group session will also be recorded using a digital audio recorder and will be transcribed in whole or in part. Transcribed names will be removed, instead being replaced by their assigned speaker numbers.

Subjects

Potential focus group participants will have to meet all of the following criteria:

* Have a diagnosis of inflammatory arthritis from a physician
* Be able to participate in a 1 ½- 2 hour focus group session
* Be aged 18 years or older
* Be English-speaking
* Be able to get to the focus group session

Recruitment and Consent Potential research participants will be identified through the Rheumatology clinics at the Sunnybrook Health Science Centre (SHSC). They will be approached by Dr. Mary Bell (Principal Investigator), staff Rheumatologist, who will introduce the study to eligible individuals and obtain their verbal consent to be contacted by the medical student co-investigator assigned to the project. The name of the individual will then be forwarded to the Office Manager who will schedule an interview at the Rheumatology clinic. At the interview, medical students will go over an information letter on the study and a consent form with each eligible patient to ensure that the potential research participant understands the study and what he/she is being asked to do. Once written consent is obtained, a copy will be provided to the participant. A confirmation letter (Appendix 4 - Confirmation Letter to Research Participants) with time and location of the interview/focus group will be mailed to the participant. The day before the interview is scheduled to take place the medical student will telephone the individual to remind them of the time and location of the interview using a Telephone Script (Appendix 5 - Telephone Script to Confirm Interview). At the beginning of the interview, prior to asking any questions, the medical student will obtain written consent and answer any further questions the participants may have.

DATA ANALYSIS

Transcripts will be analyzed using content analysis in order to systematically make inferences from text. Interview data will be imported into a NVIV0 8 qualitative software package and analyzed using a constant comparative method by the two research team members who were present at the focus group discussions. Medical students will be trained in qualitative content analysis. Interview data will be categorized into themes by each team member independently using an iterative coding scheme developed by the team. To ensure consistency in coding, the research team members who completed the focus group will frequently meet with the Principle Investigator and study coordinator to ensure consistency in coding and to verify the credibility of the codes. New codes will be added as themes arise from the data analysis. The individuals who conducted the focus group will independently code transcripts and subsequently meet compare results of the coding and agree upon their understanding of themes that emerged. By doing this cross-referencing, the rigor of the study will be increased. Modifications will be made to the interview guide with subsequent interviews to include new questions or probes that came up with prior focus group discussions. Field notes will also be used to inform the analysis.

RISKS AND BENEFITS

There are no known risks that may be associated with this study. Participants may become upset or emotional during the focus group session because the nature of the discussions will require open, honest sharing. The research team will make available a list of support groups and help-lines and reinforce that care of participants will not be affected in any way should an individual decide to withdraw from the study.

These group discussions will benefit participants as they share and discover other individuals who can relate to their disease experiences. Individuals with arthritis in Ontario may indirectly benefit in the event that this research helps develop a peer support intervention for individuals with inflammatory arthritis that may be implemented as part of the patient care process. The results of this study may help validate the importance of support based on experiential knowledge in decision-making, health promotion, and education and may encourage the implementation of peer support groups among individuals living with inflammatory arthritis.

PRIVACY AND CONFIDENTIALITY

Only the Principal Investigator, Office Manager and the medical students/study coordinator who conduct the focus group sessions will be aware of the identity of participants. All data collection forms will have identifying information removed and replaced with a unique identifying number. A list of participant names, addresses, and phone numbers will be kept on a password protected computer on a secure server in a locked research room at the rheumatology clinic at Sunnybrook Health Sciences Centre to be accessed only by the Principle Investigator and research team involved in this study. Names or other identifying information will not be used in any publications, reports, or presentations and will not be passed on to anyone else outside of the research team for this study. All information collected during the focus group sessions will be kept confidential. Hard copies of data and will be locked in a research room at Sunnybrook Health Sciences Centre for storage for 25 years before being destroyed. All electronic data files (i.e., audiofiles, transcripts) will be stored on a password protected computer on a secure server in a locked office at the Sunnybrook Health Sciences Centre rheumatology clinic. A confidentiality agreement will be signed by the study coordinator and all second year medical students involved with the study.

COMMUNICATION OF RESULTS

In terms of reporting study results, a written report will be created and sent to any participants involved in the study upon their request. A copy will also be submitted to the University of Toronto DOCH-2 Course Coordinator and the results of this study may also be shared with scientific publications, conferences, and presentations.

TEAM

Principal Investigator Mary J Bell

Co-Investigators Joyce Nyhof Young Romy Cho Chris Tran Lopamudra Das Phedias Diamandis Paula Veinot

Study Coordinator Paula Veinot

Research Assistant Gaya Embuldeniya

ELIGIBILITY:
Inclusion Criteria:

* Patients for focus groups:

  1. Have a diagnosis of IA from a physician;
  2. Able to participate in a one to two hour focus group session;
  3. 18 years of age or older;
  4. English-speaking; and,
  5. Able to get to the focus group session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory arthritis
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
learning needs (informational needs and educational preferences) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Division of Reumatology
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] REFERENCES Combe B, Landewe R , Lukas C, Bolosiu HD, Breedveld F, Dougados M et al. EULAR recommendations for the management of early arthritis: report of a task force of the European Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2007 Jan;66(1):34-45. Epub 2006 Jan 5. Dennis CL. Peer support within a health care context: A concept analysis. International Journal of Nursing Studies. 2003, 40: 321-32. Doull M, O'Connor AM, Robinson V, Tugwell P, Wells GA. Peer support strategies for improving the health and well-being of individuals with chronic diseases. (Protocol) Cochrane Database of Systematic Reviews 2005, Issue 3. Art. No.: CD005352. DOI: 10.1002/14651858.CD005352. Hunsche E, Chancellor JVM, Bruce N, The burden of arthritis and nonsteroidal anti-inflammatory treatment. A European literature review. Pharmacoeconomics. 2001;19 Suppl (1):1-15. Holbrook AM. Ontario treatment guidelines for osteoarthritis, rheumatoid arthritis, and acute musculoskeletal injury. Toronto (ON): Queen's Printer of Ontario, 2000. Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, et al. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003, 62(12):1145-55. Keysor, J. J., DeVellis, B. M., DeFriese, G. H., DeVellis, R. F., Jordan, J. M., Konrad, T. R. et al. (2003). Critical review of arthritis self-management strategy use. Arthritis Rheum. 2003, 49:724-731. Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. Perruccio AV, Power JD, Badley EM. Revisiting arthritis prevalence projections--it's more than just the aging of the population. J Rheumatol. 2006, 33(9):1856-62.